CLINICAL TRIAL: NCT00579189
Title: Safety and Efficacy of a Topical Otic Formulation in the Treatment of Acute Otitis Media With Otorrhea Through Tympanostomy Tubes (AOMT)
Brief Title: Phase III Study of an Otic Formulation in Acute Otitis Media With Tympanostomy Tubes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-05-36
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Acute Otitis Media
Keywords: ear tubes; ear drainage; ear infection; ear drops
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxidex (Experimental): Moxidex otic solution
  Interventions: Drug: Moxidex otic solution; Device: Tympanostomy tubes
- Moxifloxacin (Active Comparator): Moxifloxacin otic solution
  Interventions: Drug: Moxifloxacin otic solution; Device: Tympanostomy tubes

INTERVENTIONS:
Drug: Moxidex otic solution — 4 drops into the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxidex
Drug: Moxifloxacin otic solution — 4 drops into the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxifloxacin
Device: Tympanostomy tubes — Tubes surgically inserted through the ear drum for the treatment of recurrent otitis media in children

SUMMARY:
The purpose of this study is to determine if a topical otic formulation is safe and effective in treating middle ear infections in patients with ear tubes.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 12 years old
* Ear tubes in one or both ears
* Ear drainage visible by the parent / guardian
* Ear drainage less than 21 days
* Ear tube may not be silver oxide, silver salt, t-type tube or long-shafted tube
* Patient may not have non-tube otorrhea
* Patient may not have had otic surgery other than tube placement in the last year
* Patient may not be a menarchal female
* Diabetic patients are not eligible
* Patient may not have any disease or condition that would negatively affect the conduct of the study
* Patient may not require any other systemic antimicrobial therapy during the study.
* Patient must meet certain medication washouts to be eligible
* Analgesic use (other than acetaminophen) is not allowed
* Patient may not be pre-disposed to neurosensory hearing loss
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Age
* Other protocol-defined exclusion criteria may apply

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 776 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time to cessation of otorrhea as recorded by the parent or guardian via a patient diary | From baseline

SECONDARY OUTCOMES:
Clinical cure rate | From baseline
Microbiological outcome | From baseline
Treatment failures | From baseline

CONTACTS AND LOCATIONS:
Overall Officials: Contact Alcon Call Center, Study Director — 1-888-451-3937